CLINICAL TRIAL: NCT03290404
Title: Descriptive Assessment of Practice in Anaesthesia : Lidocaine 1% Adrenaline Under in Axillary Block Realization
Acronym: fLACON
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC17.0072 fLACON
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2017-11

CONDITIONS: Axillary Block
Keywords: Axillary Block; LidocaÏne 1% adrenaliné

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Axillary block is the good anesthetic technique for upper limb surgery without exceeding a certain total dose injected of Local Anesthetic (AL).

The maximal recommended dose of Lidocaine adrenaline in the upper limb is 500 mg. The use of ultrasound helps guiding the locoregional anesthesia, and allows to decrease the AL concentration, thus decreasing the risks.

No previous study estimated a concentration of lidocaine lower than 1,5 % to realize upper limb surgery by axillary block.

The literature overestimating probably the rate of failure of the locoregional anesthesia under ultrasound-guidance, we suggest to estimate the rate of failure of the axillary block ultrasound-guided with the lidocaine 1 % adrenaline for realizing upper limb surgery in standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for the upper limb under block axillaire
* Adult
* non-opposition

Exclusion Criteria:

* medical advice to realize axillary block
* medical advice to local anaesthetic
* Allergy
* Pregnant
* ASA 3 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult operated for the upper limb under block axillaire
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Resort to an anesthesia for help in case of ineffectiveness of the block | Day 1
  Yes or no Yes or No

SECONDARY OUTCOMES:
Block depth | Day 1
  Bromage score

OTHER OUTCOMES:
Time of Block | Day 1
  Minutes
Total dose of Lidocaïne adrenaline used | Day 1
  mg
Patient satisfaction | Day 1
  questionnaire score

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Instruction des Armées, Brest
  - CHRU de Brest, Brest
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper